CLINICAL TRIAL: NCT01979003
Title: A Pilot Study to Determine the Efficacy of Fluorescein Visualization of the Uterus in Detecting Endometrial Cancer Invasion
Brief Title: Efficacy of Fluorescein Visualization of the Uterus in Detecting Endometrial Cancer Invasion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202459
Record Dates: First submitted 2013-10-18; First posted 2013-11-08 (Estimated); Results first posted 2021-12-10 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-11

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluorescein Injection (Experimental): All research participants will receive fluorescein injection through existing intravenous line during the operative procedure. This will consist of one ampule (5 cc) injected intravenously 5- 10 minutes prior to ligation of the uterine arteries.
  Interventions: Drug: Fluorescein

INTERVENTIONS:
Drug: Fluorescein

SUMMARY:
To determine if Fluorescein systemic injection during hysterectomy procedure can be useful in revealing the depth of endometrial cancer invasion.

DETAILED DESCRIPTION:
All research participants will receive fluorescein injection through their existing intravenous line during their operative procedure for endometrial cancer staging. This will consist of one ampule (5 cc) injected intravenously prior to ligation of the uterine arteries. After the uterus is removed it will be sent to surgical pathology for evaluation as per routine care. The pathologist will open the uterus and evaluate the endometrium. He or she will then cut into the myometrium in an area most suspicious for invasion. The cross section of the myometrium and endometrium will be photographed while exposed to a Woods lamp. The normal myometrium will have a yellow fluorescent appearance under the Woods lamp. The cancerous tissue will have minimal fluorescence. The measurement will be taken estimating the depth of invasion of the cancer into the myometrium on the basis of its physical appearance under the Woods lamp. Cross-sectioning of the uterus is routine procedure by pathology for the intra-operative evaluation of endometrial cancer. This information routinely is provided in order to determine if lymph node staging is necessary.

The area that was measured and photographed will then be prepared for a frozen section to document depth of invasion. This is the standard procedure performed during an endometrial staging. The depth of invasion on the frozen section will be recorded. This same area will undergo histologic confirmation by permanent pathology to determine depth of invasion. The frozen section is part of routine standard of care in evaluation of endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Documented endometrial cancer and scheduled for hysterectomy as part of their treatment.
* No known allergy to fluorescein dye
* Ability to understand and sign informed consent
* 18 years of age or older

Exclusion Criteria:

* Prior hysterectomy
* Known sensitivity to fluorescein dye

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Burnett, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluorescein Injection: All research participants will receive fluorescein injection through existing intravenous line during the operative procedure. This will consist of one ampule (5 cc) injected intravenously 5- 10 minutes prior to ligation of the uterine arteries.
  Fluorescein
Period: Overall Study
Arm/Group | Fluorescein Injection
Started | 100
Completed | 72
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | Fluorescein Injection
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 37
Age, Continuous [Mean (Full Range); unit: years] | 62.53 [30 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 78
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Positive Predictive Value and Negative Predictive Value From Fluorescein Visualization
Description: Cancerous tissue will be measured to estimate the depth of invasion on the basis of physical appearance after receiving fluorescein injection prior to surgery. For each study subject, the paired difference in invasion depths determined using the Systemic Fluorescein Injection (SFI) versus Frozen Section (FS) methods will be calculated and expressed as a percentage of the FS-based invasion depth.
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Arm/Group | Fluorescein Injection
Number analyzed (Participants) | 72
percentage of participants
  Fluorescein Positive Predictive Value | 71
  Frozen section Positive Predictive Value | 100
  Fluorescein Negative Predictive Value | 85
  Frozen section Negative Predictive Value | 90

ADVERSE EVENTS:
Time Frame: On day of assessment.
Arm/Group | Fluorescein Injection
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

LIMITATIONS AND CAVEATS:
The protocol was updated and the other outcome measures are no longer part of the study, so they were removed. Deleted outcome measures were not pre-specified primary or secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT01979003/Prot_SAP_000.pdf